CLINICAL TRIAL: NCT00071552
Title: Evaluation of Clinical Efficacy of HFA-Propelled Beclomethasone Dipropionate Metered-Dose Inhaler Versus Fluticasone Propionate Multidose Dry Powder Inhaler on Small Airways in Poorly Controlled Asthmatic Adolescent and Adult Patients
Brief Title: Efficacy of QVAR vs Flovent Diskus on Small Airways in Poorly Controlled Asthmatic Adolescents/Adult Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Very poor enrollment
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IXR-402-4-196
Record Dates: First submitted 2003-10-28; First posted 2003-10-29 (Estimated); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Asthma
Keywords: Poorly Controlled Asthma
MeSH Terms: conditions — Asthma | interventions — Beclomethasone; Fluticasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Qvar (Experimental): Qvar 160 mcg twice daily
  Interventions: Drug: Qvar
- Flovent Diskus (Active Comparator): Flovent Diskus 200 mcg twice daily
  Interventions: Drug: Flovent Diskus

INTERVENTIONS:
Drug: Qvar — Qvar (HFA-propelled beclomethasone dipropionate metered dose inhaler) 160 mcg twice daily for 12 weeks
  Arms: Qvar
Drug: Flovent Diskus — Flovent Diskus (fluticasone propionate multi-dose dry powder inhaler) 200 mcg twice daily for 12 weeks
  Arms: Flovent Diskus

SUMMARY:
The primary objective of this study is to evaluate the effect of Beclomethasone dipropionate HFA on small airways compared to Fluticasone propionate powder for inhalation administered twice daily to poorly controlled asthmatics.

ELIGIBILITY:
Inclusion Criteria:

* Poorly controlled asthma;
* Average use of over 2 puffs of albuterol per day in the previous 7 days OR Having symptoms of asthma on 5 of the last 7 days OR Awakening at night due to asthma at least once in the previous 7 days OR Having been treated with a course of oral or intravenous steroids at least once in the last 3 months.

Exclusion Criteria:

* Subjects receiving escalating doses of immunotherapy, oral immunotherapy or short course (rush) immunotherapy for rhinitis;
* Requires beta-blockers, MAO inhibitors, tricyclic antidepressants, oral or intranasal anticholinergics;
* History and/or presence of any non-asthmatic acute or chronic lung disease, including but not limited to bronchitis, emphysema, active tuberculosis, bronchiectasis or cystic fibrosis;
* History and/or presence of any clinically significant cardiovascular disease, clinically significant hepatic, renal, or endocrine dysfunction, stroke, uncontrolled diabetes, hyperthyroidism, convulsive disorders, neoplastic disease other than basal cell carcinoma, and significant psychiatric disease.

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2004-01-31 (Actual); Primary Completion 2006-07-31 (Actual); Study Completion 2006-07-31 (Actual)

PRIMARY OUTCOMES:
Change in post-inhalation percent-predicted FEF 25-75 (%) from baseline (week 0) to week 12 | Final Visit

SECONDARY OUTCOMES:
Mean and mean change from pre-dose to 15-minute post-dose in percent predicted FEV1 (%) at week 12 | week 12

CONTACTS AND LOCATIONS:
Locations (1):
- National Jewish Medical and Research Center, Denver, Colorado, United States